CLINICAL TRIAL: NCT01438944
Title: Evaluation of Nicotine Receptor Up-regulation Activity Through Metabolic Induction and Changes in Responsiveness Using Surrogate Evaluation Methods
Brief Title: Evaluation of Transdermal Nicotine Replacement Therapy (NRT) Activity Through Metabolic Induction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Queen Elizabeth Hospital (Other)
Collaborators: Basil Hetzel Institute for Translational Research (Unknown); University of Adelaide (Other); University of South Australia (Other); Clinical Practice Unit (Unknown); Therapeutics Research Centre (Unknown)
Responsible Party: Principal Investigator, Kristin Carson, Trial co-ordinator, The Queen Elizabeth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011039
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Smoking; Addiction
Keywords: NRT; Patch; smoking; addiction
MeSH Terms: conditions — Smoking; Behavior, Addictive | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nicabate 21mg transdermal NRT (Other): 21mg Transdermal NRT applied for 24hrs over a 14day period.
  Interventions: Drug: Nicabate 21mg transdermal NRT

INTERVENTIONS:
Drug: Nicabate 21mg transdermal NRT — Nicabate 21mg Transdermal NRT Patch applied daily for 14 days Testing at Baseline, Day 4, Day 14 and 14 days post.
  Other Names: Nicotine replacement therapy

SUMMARY:
Evaluation to determine if auto-induction can be used as a surrogate measure of nicotine receptor up-regulation through an observational study using nicotine replacement therapy for two weeks and no intervention for two weeks.

DETAILED DESCRIPTION:
Studies have shown that prolonged exposure to nicotine reinforces addiction. The act of smoking delivers nicotine through lungs into the blood stream. As a result, during smoking nicotine levels peak and then when smoking stops levels progressively diminish to a base (trough) level. At the peak level a smoker feels rewarded, but at the trough level a smoker starts to experience negative withdrawal affects and a desire to smoke. Nicotine Gum and Inhalers mimic this smoking behaviour maintaining a peak and trough regime, but nicotine patches do not. Instead, nicotine patches deliver a constant base dose considered to be either above that of the smokers trough level or at a level where negative withdrawal effects are reduced.

The question arises as to if nicotine levels delivered by a patch are constant and potentially above that of the baseline smokers level, does this reinforce the addiction and therefore contribute to the high long term relapse rate? To answer this question the investigators will be looking at metabolites which the body uses to breakdown nicotine and several other enzymes. These metabolites respond to the levels of nicotine in the blood stream by increasing or decreasing over time. By testing blood flow, blood and urine the investigators are able to gain an insight into how the body is dealing with a constant stable dose of nicotine rather than a peak and trough dose. In combination with the questionnaires the investigators will be able to determine the level of affect.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who currently smoke at least 10 cigarettes per day
* Aged between 18 and 75
* Informed consent
* Willingness to attempt to quit smoking for the period specified, initially with a transdermal patch for 14 days and then without any smoking cessation aids for a further 14 days.

Exclusion Criteria:

* Use of bupropion, champix or nicotine containing products other than cigarettes in the last 2 months
* previous reactions to NRT
* Pregnancy / Breast Feeding
* Uncontrolled hypertension
* Unstable angina
* Heart attack or stroke within the previous 6 months
* Severe Obesity as indicated by Body Mass Index (BMI) ≥35 (potential for slow release of nicotine from tissues)
* acute psychiatric illness, past history psychosis, suicidal ideation or current diminished capacity.
* Current treatment or recent diagnosis of cancer
* Current use of Phenobarbital or other anticonvulsant drugs (induction of metabolism of nicotine to cotinine)
* Renal failure (creatinine clearance<30ml/min - reduces metabolic clearance of cotinine and nicotine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline Nicotine, cotinine, Leptin and orexin Metabolite ratios | Baseline, Day 4, Day 14 and Day 28
  Baseline Prior to Transdermal NRT patch application Day 4 NRT Patch Application Day 14 Last Day NRT Patch Application Day 28 14 Days post NRT patch removal.

SECONDARY OUTCOMES:
Change from baseline Patient Instruments: Fagerstrom Test for Nicotine Dependence (FTND), Wisconsin Smoking Withdrawal Scale (WSWS), Michigan Nicotine Reinforcement Questionnaire (MNRQ), Smoker Diary | Baseline, Day 14 and Day 28
  Comparative evaluation patient instruments with ratios of metabolite induction

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roberts, BPharm PhD, Principal Investigator — University of Queeensland, University of South Australia; Brian Smith, MBBS, PhD, Principal Investigator — Queen Elizabeth Hospital, University of Adelaide; Thomas Robertson, PhD, Principal Investigator — Therapeutics Research Centre; Micahel Ward, PhD, Principal Investigator — University of South Australia; John Beltrame, MBBS, FRACP, Principal Investigator — Queen Elizabeth Hospital, University of Adelaide; Malcolm Brinn, BHlthSc, Principal Investigator — Clinical Practice Unit; Kritin Carson, PhD, Principal Investigator — Clinical Practice Unit
Locations (1):
- Kristin Carson, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Available upon request